CLINICAL TRIAL: NCT04875689
Title: Effects of Laser Therapy on Chronic Knee Joint Osteoarthritis Patients
Brief Title: Laser Therapy on Chronic Knee Joint Osteoarthritis Patients PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Letter-00767Mahnoor Hanif
Record Dates: First submitted 2021-05-01; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Knee Osteoarthritis
Keywords: WOMAC; ROM; NPRS; OA
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental) (Experimental): Patient receive laser therapy along with conventional therapy
  Interventions: Other: Group A (Experimental
- Group B: Conventional treatment (Other): patient will receive conventional therapy
  Interventions: Diagnostic Test: Group B (Control)

INTERVENTIONS:
Other: Group A (Experimental — Laser therapy is performed on patients in supine lying position. Treatments will be delivered with a diode laser (wavelength 830 nm, continuous wave, power 50 mW) in skin contact at a dose of 6 J/point. Treatment times per point are in the range of 30 seconds to 1 minute. eight points were irradiated per session.
  Conventional therapy will include:
  * TENS for 15 minutes
  * Hot pack for 15 minutes
  * Hamstrings muscle stretching and calf muscle stretching. Strengthening exercises ,straight leg raising exercise in crook lying position
  * Joint mobilizations
  Arms: Group A (Experimental)
Diagnostic Test: Group B (Control) — 1. Participants of this group will receive only conventional therapy which will include;
  * TENS for 15 minutes
  * Hot pack for 15 minutes
  * Hamstrings muscle stretching and calf muscle stretching.Each stretch was sustained for 30 seconds, with 10-second rest intervals.
  * Strengthening exercises include quadricep drills(full knee extension maintained for 5 seconds, followed by a 5-second rest) 20 repetitions per session,straight leg raising exercise in crook lying position(the patients were asked to tense the quadriceps muscle, elevate the limb to 45° and maintain it for 6 seconds, and lower the limb slowly and then relax for 6 seconds; the exercise was performed for three sets of 10 repetitions per session).
  * Joint mobilizations (tibiofemoral extension and flexion; patellofemoral medial-lateral and inferior glide).
  Arms: Group B: Conventional treatment

SUMMARY:
Knee osteoarthritis is the most common condition presented in physiotherapy OPD.LASER therapy is new treatment option and to find out its effects in knee osteoarthritis is need of the hour. With this research one can find out best treatment program for knee osteoarthritis patients which can be shared with other community members. If there will be added effect of LASER treatment in reducing the visits or stays it will be a cost effective option. this study will help to find better management option for patients with knee osteoarthritis.

This study will address the scarcity of research on this topic in Pakistan and will help to raise awareness among patients about the effects of LASER THERAY.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative joint disease characterized by the loss of articular cartilage, subchondral bone remodeling, joint space narrowing and the formation of bone spurs. The initiation of cartilage breakdown is stimulated by mechanical stress or injury and the degenerative process progresses slowly over many years. In the advanced stage of OA, the abnormal remodeling of cartilage and subchondral bone results in the formation of osteophytes at the joint surface and margins, which irreversibly destroys the affected joint. Obesity, previous trauma, female gender and older age are considered the most common risk factors for knee OA. The prevalence of radiographic KOA for all age groups and found a value of 27.3 % for women and 21.0 % for men.Clinical manifestations include joint pain, stiffness, decreased range of motion (ROM), muscle weakness, proprioceptive changes, difficulties in activities of daily living (ADL) such as walking, climbing / descending stairs and housekeeping[5]Many physical therapy agents such as ultrasound[6], electrical stimulation, strengthening exercise[8]and thermal therapy[9] have been introduced.

Because of the non-invasiveness and advantage of inciting nearly no adverse side effects, low-level laser therapy (LLLT) has been widely used to relieve pain in different musculoskeletal disorder. It also promotes fibroblasts, collagen synthesis, cell oxygen recovery, and bone remodeling. Laser efficacy depends on 4 factors of wavelength, duration of treatment, dose, and areas of the application.Low level laser therapy induces photochemical physiological actions in living tissues at the cellular level. Some of these effects include cellular oxygenation, release of neurotransmitters associated with pain modulation and release of anti-inflammatory, endogenous mediators. LLLT consists of a monochromatic light source without any thermal effect that stimulates reparative properties in human cartilage. Moreover, it has an analgesic effect, although the mechanisms through which this occurs remain uncertain. The suggested mechanisms include: increased mitochondrial ATP and tissue oxygenation, increased levels of neurotransmitters implicated in pain modulation (such as serotonin) and anti-inflammatory effects. Study stated that the reduction in pain through using LLLT might be due to mechanisms such as physiological effects mediated by photochemical actions at cellular level in animal or human tissue, and through increased levels of the neurotransmitters implicated in pain modulation, such as serotonin. Some researchers have also concluded that LLLT has an effect on joint cartilage regeneration, achieved through proliferation of chondrocytes and synthesis and secretion of extracellular matrix.

A study on "Effect of laser therapy on chronic osteoarthritis of the knee in older subjects" showed that there was a significant reduction in VAS and pain intensity, an increase in isometric muscle strength and range of motion of the knee as well as increase in physical functional ability in three treatment groups.

A study on "Efficacy of low-level laser therapy on pain and disability in knee osteoarthritis: systematic review and meta-analysis of randomized placebo-controlled trials" showed that LLLT reduces pain and disability in KOA at 4-8 J with 785-860 nm wavelength and at 1-3 J with 904 nm wavelength per treatment spot.

A study on "effectiveness of low-level laser therapy in patients with knee osteoarthritis: a systematic review and meta-analysis" this study indicated that low level laser therapy has neither early nor later benefits in reducing pain or improving function in patients with KOA.

A study on "The Effect of Low Level Laser Therapy on Pain and Range of Motion of Patients With Knee Osteoarthritis" showed that the effectiveness of low-power laser in reducing pain and improving the range of motion in patients with knee osteoarthritis is similar to the effectiveness of the placebo laser. Low-power laser is recognized as an appropriate medical modality to treat knee osteoarthritis in animals and humans and can be used along with acupuncture or exercise.

A study on Effect of low level laser therapy (904nm) and static stretching in patients with knee osteoarthritis: a protocol of randomized controlled trial showed that the The European League Against Rheumatism (EULAR) recommendations indicate stretching exercises as an adjunctive treatment.

ELIGIBILITY:
Inclusion Criteria:

* • The study includes female patients with chronic knee OA

  * The study includes patients from the age of 40 years and 65 years
  * The study includes patients with Grade II and III OA of knee
  * Patients having no other physical and mental issues

Exclusion Criteria:

* • The study excludes male patients

  * Patients with lab results abnormal (inflammatory and infectious disease, malignant tumor)
  * Patients with arterial coagulation blockage in lower limbs.
  * Usual contraindication for laser therapy
  * Patient's undergone surgery of knee

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females
Enrollment: 42 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
WOMAC questionnaire | 12th day
  It is a self-administered questionnaire consisting of 24 items divided into 3 subscales.
  • Test-retest reliability of pain,stiffness and physical function was satisfactory with ICCs(intraclass correlation coefficients) of 0.86, 0.68, and 0.89, respectively.
Goniometry | 12th day
  knee ROM can be measured with this tool
NPRS | 12th day
  • Numeric pain rating scale: numeric pain rating scale (NPRS) is ascale for pain measurement, ranging from "0" representing no pain :10" representing the worst or severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Shafaq Shahid, MSPT(OMPT), Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral,Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JK, Kim TH, Park SW, Kim HY, Kim Sh, Lee Sy, Lee SM. Protective effects of human placenta extract on cartilage degradation in experimental osteoarthritis. Biol Pharm Bull. 2010;33(6):1004-10. doi: 10.1248/bpb.33.1004. PMID 20522967
- [Background] Blagojevic M, Jinks C, Jeffery A, Jordan KP. Risk factors for onset of osteoarthritis of the knee in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2010 Jan;18(1):24-33. doi: 10.1016/j.joca.2009.08.010. Epub 2009 Sep 2. PMID 19751691
- [Background] Pereira D, Peleteiro B, Araujo J, Branco J, Santos RA, Ramos E. The effect of osteoarthritis definition on prevalence and incidence estimates: a systematic review. Osteoarthritis Cartilage. 2011 Nov;19(11):1270-85. doi: 10.1016/j.joca.2011.08.009. Epub 2011 Aug 24. PMID 21907813
- [Background] Kaufman KR, Hughes C, Morrey BF, Morrey M, An KN. Gait characteristics of patients with knee osteoarthritis. J Biomech. 2001 Jul;34(7):907-15. doi: 10.1016/s0021-9290(01)00036-7. PMID 11410174
- [Background] Bennell KL, Hunt MA, Wrigley TV, Hunter DJ, Hinman RS. The effects of hip muscle strengthening on knee load, pain, and function in people with knee osteoarthritis: a protocol for a randomised, single-blind controlled trial. BMC Musculoskelet Disord. 2007 Dec 7;8:121. doi: 10.1186/1471-2474-8-121. PMID 18067658
- [Background] Zeng C, Li H, Yang T, Deng ZH, Yang Y, Zhang Y, Ding X, Lei GH. Effectiveness of continuous and pulsed ultrasound for the management of knee osteoarthritis: a systematic review and network meta-analysis. Osteoarthritis Cartilage. 2014 Aug;22(8):1090-9. doi: 10.1016/j.joca.2014.06.028. Epub 2014 Jul 4. PMID 24999112
- [Background] Melo Mde O, Pompeo KD, Brodt GA, Baroni BM, da Silva Junior DP, Vaz MA. Effects of neuromuscular electrical stimulation and low-level laser therapy on the muscle architecture and functional capacity in elderly patients with knee osteoarthritis: a randomized controlled trial. Clin Rehabil. 2015 Jun;29(6):570-80. doi: 10.1177/0269215514552082. Epub 2014 Sep 26. PMID 25261425
- [Background] Uthman OA, van der Windt DA, Jordan JL, Dziedzic KS, Healey EL, Peat GM, Foster NE. Exercise for lower limb osteoarthritis: systematic review incorporating trial sequential analysis and network meta-analysis. BMJ. 2013 Sep 20;347:f5555. doi: 10.1136/bmj.f5555. PMID 24055922
- [Background] Huang Z, Chen J, Ma J, Shen B, Pei F, Kraus VB. Effectiveness of low-level laser therapy in patients with knee osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Sep;23(9):1437-1444. doi: 10.1016/j.joca.2015.04.005. Epub 2015 Apr 23. PMID 25914044
- [Background] Coelho Cde F, Leal-Junior EC, Biasotto-Gonzalez DA, Bley AS, de Carvalho Pde T, Politti F, Gonzalez Tde O, de Oliveira AR, Frigero M, Garcia MB, Dibai-Filho AV, Gomes CA. Effectiveness of phototherapy incorporated into an exercise program for osteoarthritis of the knee: study protocol for a randomized controlled trial. Trials. 2014 Jun 11;15:221. doi: 10.1186/1745-6215-15-221. PMID 24919587
- [Background] Al Rashoud AS, Abboud RJ, Wang W, Wigderowitz C. Efficacy of low-level laser therapy applied at acupuncture points in knee osteoarthritis: a randomised double-blind comparative trial. Physiotherapy. 2014 Sep;100(3):242-8. doi: 10.1016/j.physio.2013.09.007. Epub 2013 Nov 15. PMID 24418801